CLINICAL TRIAL: NCT06244992
Title: A Phase 1/2a Study to Evaluate the Safety, Pharmacokinetics and Efficacy of PTT-936, an Alpha Kinase 1 (ALPK1) Activator, Alone or in Combination With Anti-PD-1/L1 in Patients With Locally Advanced or Metastatic Solid Tumors
Brief Title: PTT-936 Alone or in Combination in Patients With Locally Advanced or Metastatic Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Pyrotech Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PTT-936-101
Record Dates: First submitted 2024-01-16; First posted 2024-02-06 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Locally Advanced or Metastatic Solid Tumors
Keywords: Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- PTT-936 Dose Level 1 (Experimental): PTT-936 will be administered once a week (QW)
  Interventions: Drug: PTT-936
- PTT-936 Dose Level 2 (Experimental): PTT-936 will be administered once a week (QW)
  Interventions: Drug: PTT-936
- PTT-936 Dose Level 3 (Experimental): PTT-936 will be administered once a week (QW)
  Interventions: Drug: PTT-936
- PTT-936 Dose Level 4 (Experimental): PTT-936 will be administered once a week (QW)
  Interventions: Drug: PTT-936
- PTT-936 Dose Level 5 (Experimental): PTT-936 will be administered once a week (QW)
  Interventions: Drug: PTT-936
- PTT-936 and anti-PD-1/L1 combination therapy (Experimental): PTT-936 will be administered once a week (QW) in combination with a standard-of-care (SOC) regimen of an anti-PD-1/L1 agent every three weeks (Q3W)
  Interventions: Drug: Combination of PTT-936 and anti-PD-1/L1 therapy

INTERVENTIONS:
Drug: PTT-936 — Eligible patients will receive single-agent PTT-936 administered per orally (PO).
  Arms: PTT-936 Dose Level 1; PTT-936 Dose Level 2; PTT-936 Dose Level 3; PTT-936 Dose Level 4; PTT-936 Dose Level 5
Drug: Combination of PTT-936 and anti-PD-1/L1 therapy — Eligible patients will receive combination treatment consisting of PTT-936 administered PO in combination with a Standard of Care (SOC) regimen of an anti-PD-1/L1 agent administered intravenously (IV).
  Arms: PTT-936 and anti-PD-1/L1 combination therapy

SUMMARY:
This Phase 1/2a study will explore the safety and efficacy of PTT-936, an Alpha Kinase 1 (ALPK1) activator, used alone or in combination with anti-PD-1/L1 therapy in patients with locally advanced or metastatic solid tumors. The study is divided into two parts: Phase 1 (Part A) focuses on determining the pharmaceutically active dosage range and evaluating the safety profile of PTT-936 when administered as a monotherapy. Phase 2a (Part B) will assess the safety and efficacy of PTT-936 combined with anti-PD-1/L1 therapy in patients suitable for anti- PD-1/L1 monotherapy. The study aims to understand how PTT-936, alone or in combination, impacts tumor progression and patients' overall response.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily signed informed consent form (ICF).
2. Ability and willingness to adhere to all study procedures.
3. Male or female patients ≥ 18 years of age at the time of signing the ICF.
4. Locally advanced unresectable or metastatic solid tumor confirmed by histology or cytology
5. For Part A: On tumor imaging, as assessed by RECIST v1.1 and iRECIST, with measurable or unmeasurable disease. For Part B: On tumor imaging, as assessed by RECIST v1.1 and iRECIST, with at least one measurable disease.
6. Life expectancy ≥ 3 months.
7. Eastern Cooperative Oncology Group (ECOG) performance status (PS): 0-1 for Part A and Part B.
8. Adequate end-organ and hematopoietic function, defined based on the following laboratory results obtained within 7 days prior to the first dose of study treatment [Day 1]):

   1. Absolute neutrophil count (ANC) ≥ 1.5×109/L (1500/μL), without granulocyte colony-stimulating factor (G-CSF) support. Note that G-CSF may be administered until 14 days prior to Cycle 1 Day 1 (C1D1).
   2. Platelet count ≥ 90×109/L (90,000/μL) without transfusion within 14 days prior to C1D1.
   3. Hemoglobin ≥ 90 g/L (9 g/dL). Note that patients may be transfused or receive erythropoietic treatment to meet this criterion until 14 days prior to C1D1.
   4. Creatinine clearance ≥ 60 mL/min.
   5. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 3 x the upper limit of normal (ULN) with or without primary or metastatic liver tumor lesions.
   6. Total bilirubin (TBIL) ≤ 1.5 x ULN.
   7. For patients not receiving therapeutic anticoagulation: International Normalized Ratio (INR), activated partial thromboplastin time (aPTT) and prothrombin time (PT) ≤ 1.5 x ULN.
   8. For patients receiving warfarin: INR ≤ 3.0 x ULN and no bleeding within 14 days prior to Day 1. Patients receiving therapeutic anticoagulation must be on a stable dose for a minimum of 14 days prior to Day 1. Patients on low molecular weight heparin will be allowed.

Exclusion Criteria:

1. Patients with leptomeningeal (LMD) metastases or patients with new and/or progressive brain metastases at the time of study entry. Patients with treated brain metastases are eligible if there is no evidence of progression for at least 4 weeks after central nervous system (CNS)-directed treatment (radiotherapy and/or surgery), as ascertained by clinical examination and brain imaging (MRI or CT) during the screening period.
2. History of primary malignancy other than the diseases under study, not in remission greater than three (3) years prior to Day 1. Exceptions that do not require a 3-year remission include: adequately treated non-melanoma skin cancer, cervical carcinoma in situ on biopsy or squamous intraepithelial lesion on Papanicolaou (PAP) smear, in situ prostate cancer (with no evidence of active disease for two [2] years prior to Day 1), or resected melanoma in situ and radically resected papillary thyroid carcinoma.
3. Persistence of Adverse Events (AEs) from prior anti-cancer therapy that have not resolved to Grade 1 (except for alopecia and hypothyroidism), or any history of Grade ≥ 3 immune-related adverse events (irAEs), Grade ≥ 2 pneumonitis, hypophysitis or encephalitis related to immunotherapy, or other Grade ≥ 3 drug-related CNS toxicity.
4. Active systemic autoimmune disease or a history of autoimmune disorder that may relapse (e.g., systemic lupus erythematosus [SLE], rheumatoid arthritis, inflammatory bowel disease [IBD], autoimmune thyroid disorder*, multiple sclerosis, vasculitis, glomerulitis, eczema, psoriasis, etc.).

   *Note that primary or secondary hypothyroidism, well controlled with hormone replacement therapy is permitted.
5. Major trauma or major surgery within 4 weeks prior to Day 1 or anticipated major surgery during study participation.
6. Serious unhealing wound, ulcer, or bone fracture.
7. History of and/or presence of any of the following cardiovascular and cerebrovascular events or conditions:

   1. History of myocardial infarction, unstable or severe angina, or arterial thrombotic event (such as cerebrovascular attack [CVA] or transient ischemic attack [TIA]) within 12 months prior to Day 1.
   2. Significant abnormalities on the screening of ECG, including corrected QT interval (QTc interval) > 470 msec (average of triplicate measurements, corrected for heart rate using Fridericia's formula), second degree (Mobitz type II) or third degree atrioventricular (AV) block, or other clinically significant (in the Investigator's opinion) arrhythmia.
   3. Current New York Heart Association (NYHA) stage II-IV congestive heart failure (CHF).
   4. Left ventricular ejection fraction (LVEF) < 50%.

      • Note that LVEF assessment by echocardiogram (ECHO) scan performed as part of the patient's regular care within 4 weeks prior to the screening visit may be used for confirmation of eligibility.
   5. Other clinically significant (in the Investigator's opinion) cardiac diseases (e.g., valvular disease, cardiomegaly, ventricular hypertrophy, cardiomyopathy, myocarditis, etc.).
   6. Uncontrolled hypertension (defined as a systolic blood pressure [SBP] ≥ 150 mmHg and/or diastolic blood pressure (DBP) ≥ 100 mmHg at screening), despite appropriate antihypertensive therapy, or poor compliance with an antihypertensive regimen.
8. Active or recent (past 6 months) bleeding disorder, including gastrointestinal (GI) bleeding, as evidenced by hematemesis, significant hemoptysis, or melena within 6 months prior to Day 1.
9. Uncontrolled diabetes.
10. Chronic severe liver disease or Child-Pugh B or C liver cirrhosis.
11. History of alcoholism or drug abuse within the past year.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2024-01-26 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Incidence of TEAEs and TRAEs (with severity determined using NCI CTCAE v5.0), Grade >3 TEAEs, Grade >3 TRAEs, SAEs, and AESIs | 7 months
Overall Response Rate (ORR): defined as the percentage of patients who achieved Complete Response (CR) or Partial Response (PR) according to RECIST v1.1 and iRECIST during the study | 7 months

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Precision NextGen Oncology and Research Center, Beverly Hills, California
  - D&H Cancer Research Center, Margate, Florida
  - The START Center, San Antonio, Texas